CLINICAL TRIAL: NCT03840564
Title: Impact of Biological Point of Care Devices Implementation on the Length of Stay of Patients in Emergency Room
Acronym: SUPOC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI16022HLJ
Record Dates: First submitted 2018-05-29; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-05

CONDITIONS: Emergencies; Care
MeSH Terms: conditions — Emergencies | interventions — Point-of-Care Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group point of care (POC): All the analyzes will be done in delocalized
  Interventions: Other: Point of care (POC)
- control group: the analyzes will be done at the central laboratory

INTERVENTIONS:
Other: Point of care (POC) — All the analyzes will be done in delocalized
  Groups: Group point of care (POC)

SUMMARY:
"Main objective: to demonstrate that the implementation of an extended panel solution for the point of care analysis of biological parameters (point of care : POC) in an emergency department (ED) reduces the length of stay (LOS) of patients Secondary objectives: to demonstrate the feasibility of implementing an expanded panel of POC solutions in an ED and the reduction of emergency overcrowding in the POC group.

To determine the medico-economic impact of the extended implementation of POC solutions (cost-efficiency and health-economic study), to collect the satisfaction of medical (emergency physicians, medical biologists) and paramedical personnel as well as the satisfaction of patients.

Inclusion criteria: Any patient consulting in the emergency department during the study period Non-inclusion criteria: Patients attending the emergency departments as part of dressing or trauma follow-up consultations Main criteria of judgment: Time between administrative registration and the patient's discharge or hospitalization decision, compared between the control period and the intervention period (POC).

Design: Prospective, monocentric, controlled, cluster- randomized per week. Duration of center preparation (technical preparation and training of laboratory staff): 4 weeks Duration of inclusion period: 18 weeks Duration of patient participation: 1 day Total trial duration time: 22 weeks"

DETAILED DESCRIPTION:
"SUPOC is a monocentric, prospective, open-label, controlled study, randomized into one-week inclusion periods, with 2 types of period: period POC (biological analysis performed as POC in a dedicated emergency room implemented with POC devices) and period control (analysis performed sent and processed in the central laboratory). Randomisation will be carried out by periods of one week (periods of a whole week 24h/24 from Monday 8am to Sunday 8 pm: control period or POC period, with a wash-out period between Sunday 08 pm and Monday 8am before each change of period (in order to limit the patients overlap on 2 periods). The entire medical care including the clinical examination, the prescriptions for additional radiological or biological examinations, requests for specialist advice, as well as the conclusion of the medical file will be left to the sole discretion of the emergency physician in charge of the patient and dictated solely by the reason for consultation and the patient evolution. The comparability of the POC and control periods will be verified, quantitatively (number of patients, average number of paramedical personnel present, the number of medical personnel being fixed) and qualitatively (triage scale applied by the triage nurses into 5 classes).

Despite the randomization of the two periods, the study type is best described as "Observational" because there is no specific intervention or health outcome at the subject level at all. The fact that blood samples are sent in the central laboratory or in the POC platform are both considered as routine medical care. No investigator assigns a specific intervention to the study participants; it is the emergency department itself which changes its internal organization (the destination of the biologic samples) every week. In conclusion, the purpose of the study is to examine the effect of a health provider intervention (POC vs central laboratory use) on a health provider outcome (mean length of stay according to the study period), and there is no health outcomes at the patient level. According to the ICMJE guidelines, this type of study should not be considered as an interventional clinical trial (http://www.icmje.org/about-icmje/faqs/clinical-trials-registration/).

For organizational reasons, 3 laboratory technicians will be recruited and trained specifically for the study. They will be in charge of biological testing during POC periods.

Primary evaluation criteria: length of stay (LOS) of patients consulting the ED, defined by the time between the administrative registration and the medical decision of discharge or hospitalization of the patient. This LOS for each patient meeting the eligibility criteria will be extracted by the hospital's informatic department from the emergency file database. Secondary endpoints: - -the feasibility of an expanded POC menu in the ED will be assessed by the ""converted"" analysis rate, i.e. the number of analyses sent to the central laboratory in the POC period divided by the total number of analyses performed as POC during the period, the rate of unavailability of each POC device for maintenance or breakdown, i.e. the cumulative number of minutes of unavailability for all the POC equipment compared to the total duration of the POC group's periods.

ED's crowding will be evaluated by: the waiting time in each period (time in minutes between emergency registration and first medical contact), the occupancy rate defined by - at time t- the number of patients present / ED's capacity. The capacity of the service is estimated on the basis of the total number of boxes and beds, including short-term hospitalisation units. An overcrowding is set to an occupancy rate> 150%. In practice,it will be extracted by the informatic department from emergency database every day of the study at 12pm, 6pm, 12am and 8am.

The time to results in each period and by biological parameter will be extracted from the laboratory software.

The health-economic impact of the expanded implementation of POC will be assessed by the average total cost of an ED's visit in each period. The costs and consequences of the implementation of the POC will be estimated in a comparative way in the two periods, taking into account on the one hand the point of view of the establishment and on the other hand that of the healthcare system. The investigators will estimate an average cost per patient and per emergency room visit.

The satisfaction of staff and patients will be evaluated by an anonymous questionnaire including satisfaction scales on the overall quality of care in emergency department and on the results of biological analyses, among patients (on a sample) and all staff (emergency physicians and biologists, ED's nurses).

Sample size calculation: This is a one-week randomized cluster study. A preliminary study of the first 6 months of 2016, using ED's software to extract data from emergency department visits, estimated an average cluster size of 1100 patients, with a size variation coefficient of 0.2, as well as a standard deviation of 2 hours and 20 minutes.

Assuming an average reduction of 20 minutes of the main judgement criterion, and an intraclass correlation coefficient of 0.01, with a bilateral alpha equal to 5%, study will have to include 9 clusters in each period to obtain a power of 80% - 18 weeks total duration of inclusion.

For a monocentric study including all patients consulting in an adult emergency department with a total of 60,000 visits per year, each month will allow the inclusion of at least 4,400 patients.

ELIGIBILITY:
Inclusion Criteria:

* Any patient consulting in the emergency department during the study period

Exclusion Criteria:

* Patients attending the emergency departments as part of dressing or trauma follow-up consultations

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient consulting in the emergency department
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2018-10-14 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
length of stay (LOS) of patients consulting the ED | 1 Week
  length of stay (LOS) of patients consulting the ED For each patient the time frame of LOS is comprised between the admission schedule in the ED and the schedule of medical conclusion on the medical file of each patient consulting the emergency department

SECONDARY OUTCOMES:
Incidence and duration of technical adverse events encountered with the POC platform | through study completion (18 weeks)
  "converted" analysis rate, i.e. the number of analyses sent to the central laboratory in the intervention period divided by the total number of analyses performed as POC during the period, the rate of unavailability of each POC device for maintenance or breakdown, i.e. the cumulative number of minutes of unavailability for all the POC equipment compared to the total duration of the intervention group's periods
ED's crowding | 1 Week, i.e. the size of one cluster period of observation
  Mean waiting time in each period defined by the time in minutes between the emergency admission registration schedule and the first medical contact)
The time to results in each period and by biological parameter | 1 Week, i.e. the size of one cluster period of observation
  The mean time elapsed between blood sampling an result availability for the physician
health-economic impact | through study completion (18 Weeks)
  Average total cost of an ED's visit in each period. The costs and consequences of the implementation of the POC will be estimated in a comparative way in the two periods, taking into account on the one hand the point of view of the establishment and on the other hand that of the healthcare system. We will estimate an average cost per patient and per emergency room visit.
satisfaction of patients | the last two weeks of the study: one week in the intervention period (POC) and one week in the control period (usual care)
  anonymous questionnaire including satisfaction scales on the overall quality of care in emergency department and on the time to result of biological analyses, among patients (on a sample) For each of the satisfaction criteria studied, a numeric scale will be submitted to a sample of patients . The numeric scale ranges from 1 (very low satisfaction) to 10 (very high satisfaction).
satisfaction of all staff | the last two weeks of the study: one week in the intervention period (POC) and one week in the control period (usual care)
  anonymous questionnaire including satisfaction scales on the overall quality of care in emergency department and on the time to result of biological analyses, satisfaction of all staff (emergency physicians and biologists, ED's nurses). For each of the satisfaction criteria studied, a numeric scale will be submitted to all the ED personnel . The numeric scale ranges from 1 (very low satisfaction) to 10 (very high satisfaction).

CONTACTS AND LOCATIONS:
Overall Officials: HAUSFATER Pierre, Pr, MD, PhD, Principal Investigator — Pitie salpetriere hospital
Locations (1):
- Pitié Salpetriere hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hausfater P, Hajage D, Bulsei J, Canavaggio P, Lafourcade A, Paquet AL, Arock M, Durand-Zaleski I, Riou B, Oueidat N. Impact of Point-of-care Testing on Length of Stay of Patients in the Emergency Department: A Cluster-randomized Controlled Study. Acad Emerg Med. 2020 Oct;27(10):974-983. doi: 10.1111/acem.14072. Epub 2020 Jul 27. PMID 32621374